CLINICAL TRIAL: NCT01449591
Title: A Proof of Concept (PoC) Study to Evaluate the Safety, Tolerability, and Efficacy of 12 Week Administration of BFH772 Ointment in Rosacea Patients
Brief Title: Safety, Tolerability and Efficacy of BFH772 in Rosacea Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBFH772A2203
Record Dates: First submitted 2011-09-19; First posted 2011-10-10 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Erythemato-telangiectatic Rosacea
Keywords: BFH772; rosacea; erythemato-telangiectatic rosacea
MeSH Terms: conditions — Rosacea | interventions — Ointments; Benchmarking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- BFH772 (Experimental)
  Interventions: Drug: BFH772 1% ointment
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle ointment
- Metronidazole (Active Comparator)
  Interventions: Drug: Noritate® 1% cream

INTERVENTIONS:
Drug: BFH772 1% ointment
  Arms: BFH772
Drug: Vehicle ointment
  Arms: Vehicle
Drug: Noritate® 1% cream
  Arms: Metronidazole

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of BFH772 after 12 weeks of treatment as compared to an active control and vehicle in patients with erythemato-telangiectatic rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Have persistent facial erythema on the cheeks of at least moderate severity.
* Women must not be able to bear children

Exclusion Criteria:

* Have more than 12 inflammatory lesions on the face
* Previous treatment of facial skin with lasers or electrocauterisation within 2 months prior to entering the study
* Have facial hair that makes it difficult to evaluate rosacea on the face Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess the effect of BFH772 treatment compared to vehicle on non-transient facial erythema using the Investigator's assessment of facial erythema score | 12 weeks

SECONDARY OUTCOMES:
To evaluate a patient's assessment of flushing frequency via patient reported episodes and facial redness via a patient reported score | 12 weeks
To measure blood levels of BFH772 in patients | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Paramus, New Jersey
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Spokane, Washington

REFERENCES:
- See also: Results for CBFH772A2203 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=7963